CLINICAL TRIAL: NCT06432712
Title: Comparison of Post Operative Endodontic Pain in Patients with Irreversible Pulpitis Treated with and Without Dexamethasone.
Status: Not yet recruiting | Phase: Early Phase 1 | Type: Interventional
Sponsor: Shoaib Rahim (Other)
Collaborators: Foundation University Islamabad (Other)
Responsible Party: Sponsor-Investigator, Shoaib Rahim, Assistant professor, Foundation University Islamabad
Organization: Foundation University Islamabad (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: FUCDCLINIC-2404
Record Dates: First submitted 2024-05-23; First posted 2024-05-29 (Actual); Last update posted 2024-12-13 (Actual); Status verified 2024-05

CONDITIONS: Pain
Keywords: Postoperative Pain; Root canal therapy; Dexamethasone; Pulpitis
MeSH Terms: conditions — Pain; Pain, Postoperative; Pulpitis | interventions — Dexamethasone

STUDY DESIGN:
Intervention Model Description: This is a single-blind, randomized parallel-arm study with two arms. Participants will be randomly assigned to either receive dexamethasone infiltration or only analgesic therapy. They will remain in their assigned group throughout the study.
Masking Description: Interventional or control group will be selected randomly through sealed envelope by an independent researcher not involved in the study.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Control (No Intervention): Participants in this arm will receive routine root canal treatment with a prescription of NSAIDs post operatively.
- Experimental (Experimental): Participants in this arm will receive routine root canal treatment along with 2.5ml of dexamethasone 4mg/ml peri apical infiltration with a prescription of NSAIDs post operatively.
  Interventions: Drug: Dexamethasone 4mg

INTERVENTIONS:
Drug: Dexamethasone 4mg — 2.5ml of Dexamethasone 4mg/ml will be administered via periapical infiltration with a 23 gauge needle to the experimental group.
  Arms: Experimental

SUMMARY:
Root canal procedure is a common procedure in dentistry. Acute inflammatory response in peri-radicular tissues after root canal treatment is the main cause of post op pain.

Potential Solution: The current study will assess effect of dexamethasone administered as periapical infiltration in reducing post-instrumentation pain.

Research Goal: Pain score of patients treated with dexamethasone infiltration will be less compared to patients treated with NSAIDS alone after canal instrumentation.

DETAILED DESCRIPTION:
Acute inflammatory response in peri-radicular tissues after root canal treatment is the main cause of post op pain. The peak inflammatory response occurs after 24 - 48 hours of root canal instrumentation. As management of post-endodontic pain is still a challenge for clinicians several drugs which include NSAIDs, acetaminophen, opioids and steroids are used to reduce the inflammatory response. Corticosteroids possess anti-inflammatory efficacy, and they prevent the production and release of inflammatory mediators at the site of tissue injury thus reducing the signs & symptoms of inflammation such as pain, swelling & loss of function. Dexamethasone is a potent corticosteroid that has the ability to reduce the production of proinflammatory cytokines. Dexamethasone can be administered orally, or as an intraosseous, intra ligament periapical & intracanal injection. Dexamethasone is effective in alleviating pain in first 24 hours post endodontic treatment. Previous research on the effect of dexamethasone injection on post-endodontic treatment pain in patients presenting with necrotic pulp treated with single visit endodontic treatment reported 25% post operative pain occurrence and 9% when treated with dexamethasone.

Study Goal : The current study will assess effect of dexamethasone administered as periapical infiltration in reducing post-instrumentation pain as compared to the prescription of NSAIDs only. If dexamethasone infiltration is effective in pain relief after endodontic treatment, it can be a useful adjunct in managing patients presenting with acute pulpal pain.

ELIGIBILITY:
Inclusion Criteria:

* Patients of age 18-50 years
* Maxillary molar and premolar teeth
* Pt diagnosed with irreversible pulpitis with or without apical periodontitis

Exclusion Criteria:

* Teeth with calcified canals.
* Teeth with incompletely formed apices.
* Teeth requiring retreatment.
* Taking analgesics, anti-inflammatory, or tri-cyclic anti-depressants for their medical conditions.
* Teeth with grade II or III mobility (more than 2 mm)
* Pregnant patients
* Pt who are immunocompromised (uncontrolled diabetes mellitus, renal impairment)

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 140 (Estimated)
Dates: Start 2025-01-10 (Estimated); Primary Completion 2025-01-10 (Estimated); Study Completion 2025-06-10 (Estimated)

PRIMARY OUTCOMES:
post operative pain | 12 hours, 24 hours and 1 week
  The patient's pain response before treatment will be recorded using visual analogue scale 0-10.Pain score of 3 and less than 3 will be categorized as no postoperative pain and score greater than 3 will be categorized as post operative pain.

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Suresh N, Nagendrababu V, Koteeswaran V, Haritha JS, Swetha SD, Varghese A, Natanasabapathy V. Effect of preoperative oral administration of steroids in comparison to an anti-inflammatory drug on postoperative pain following single-visit root canal treatment - a double-blind, randomized clinical trial. Int Endod J. 2021 Feb;54(2):198-209. doi: 10.1111/iej.13416. Epub 2020 Nov 12. PMID 32976660
- [Background] Yeganegi S, Fazelian N, Layegh Nejad MK, Manzouri L. Comparison of the Efficacy of Dexamethasone and Methylprednisolone in Infiltration Injection for Postendodontic Pain in Patients with Necrotic Pulp: A Randomized Controlled Clinical Trial. Pain Res Manag. 2022 Feb 23;2022:4163120. doi: 10.1155/2022/4163120. eCollection 2022. PMID 35251416
- [Background] Aksoy F, Ege B. The effect of pretreatment submucosal injections of tramadol and dexamethasone on post-endodontic pain in mandibular molar teeth with symptomatic irreversible pulpitis: a randomized controlled clinical trial. Int Endod J. 2020 Feb;53(2):176-185. doi: 10.1111/iej.13246. Epub 2019 Nov 28. PMID 31702056
- [Background] Nogueira BML, Silva LG, Mesquita CRM, Menezes SAF, Menezes TOA, Faria AGM, Porpino MTM. Is the Use of Dexamethasone Effective in Controlling Pain Associated with Symptomatic Irreversible Pulpitis? A Systematic Review. J Endod. 2018 May;44(5):703-710. doi: 10.1016/j.joen.2018.02.006. Epub 2018 Mar 20. PMID 29571913
- [Background] Yavari HR, Jafari F, Jamloo H, Hallaj-Nezhadi S, Jafari S. The Effect of Submucosal Injection of Corticosteroids on Pain Perception and Quality of Life after Root Canal Treatment of Teeth with Irreversible Pulpitis: A Randomized Clinical Trial. J Endod. 2019 May;45(5):477-482. doi: 10.1016/j.joen.2019.01.005. Epub 2019 Mar 23. PMID 30910353